CLINICAL TRIAL: NCT00358137
Title: Psychophysiologic Stress, Exercise, & Autonomic Control
Brief Title: Effect of Aerobic Exercise on Blood Pressure Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Richard P. Sloan, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 404; R01HL061287-04 (NIH)
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2007-12

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Blood Pressure, High
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Behavioral: Aerobic Conditioning Program
Behavioral: Strength Training Program

SUMMARY:
This study will evaluate the effect of an aerobic training program versus a strength training program on the autonomic nervous system at rest and in response to challenge.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of an aerobic exercise program versus a strength training program in altering RR interval and blood pressure variability as indices of autonomic nervous system regulation of the cardiovascular system. Subjects will be tested at rest and in response to challenge.

This study will enroll healthy, young (age 18-45) sedentary individuals at Columbia University Medical Center and St. John's University. At an initial screening visit, potential participants will be screened for exercise activity and will also undergo a test of aerobic capacity. Subjects will be eligible if they are not exercising regularly and do not exceed American Heart Association standards for average fitness (VO2max ≤ 43 and 37 ml/kg/min for men and women respectively). Exclusion criteria include current symptoms of affective disorder, psychosis, or substance abuse, current usage of psychotropic medication, and any medical condition that affected the autonomic nervous system or cardiovascular system.

Eligible participants will then be randomly assigned to 12 weeks of either an aerobic conditioning program or a strength training program. At study entry, heart rate, respiratory rate, and blood pressure will be measured; an ECG will be used to measure heart activity. Questionnaires will be completed to assess anger, tension, depression, and fatigue. Participants in the aerobic conditioning program will attend four 1-hour exercise sessions per week, which will focus on increasing cardiovascular fitness through running and other forms of aerobic exercise. The strength training program will also include four sessions per week, with the focus on increasing muscle endurance and strength. At the end of the 12-week programs, participants will begin a 4-week period of deconditioning, during which they will discontinue all exercise. Evaluations will be repeated at the end of the 12-week programs, and at the end of the 4-week deconditioning period.

ELIGIBILITY:
Inclusion Criteria:

* Average cardiorespiratory fitness level, as defined by the American Heart Association (VO2 max [maximum oxygen consumption] less than 43 ml/kg/min for men and less than 37 ml/kg/min for women)
* English speaking
* Ambulatory
* Sedentary

Exclusion Criteria:

* Use of psychotropic medications
* Past or current psychiatric disorder
* Heart disease
* High blood pressure
* Diabetes mellitus
* Neurologic disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 1997-07; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
RR inverval (RRV) and blood pressure variability at rest and in response to challenge (measured prior to exercise training and again after training and after sedentary deconditioning).

SECONDARY OUTCOMES:
Secondary outcome measures include ambulatory blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Sloan, PhD, Principal Investigator — Columbia University

REFERENCES:
- [Derived] Alex C, Lindgren M, Shapiro PA, McKinley PS, Brondolo EN, Myers MM, Zhao Y, Sloan RP. Aerobic exercise and strength training effects on cardiovascular sympathetic function in healthy adults: a randomized controlled trial. Psychosom Med. 2013 May;75(4):375-81. doi: 10.1097/PSY.0b013e3182906810. Epub 2013 Apr 29. PMID 23630307